CLINICAL TRIAL: NCT06961591
Title: Cooking Skills to Improve Long-Term Weight Loss in Young Adults With Intellectual Disabilities
Acronym: CHEF-ID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY 160822; R01HD116832 (NIH)
Record Dates: First submitted 2025-04-24; First posted 2025-05-08 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Intellectual Disability; Overweight and Obesity
Keywords: Weight Loss Maintenance; Cooking Skills; Weight loss; Down syndrome
MeSH Terms: conditions — Intellectual Disability; Overweight; Obesity; Weight Loss; Down Syndrome | interventions — Cooking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight Loss Plus Cooking (Experimental)
  Interventions: Behavioral: Weight Loss Plus Cooking
- Traditional Weight Loss (Active Comparator)
  Interventions: Behavioral: Traditional Weight Loss

INTERVENTIONS:
Behavioral: Weight Loss Plus Cooking — Participants in the eSLD+Chef-ID group will follow a healthy eating plan using the enhanced stoplight diet, meet with a health coach once a month on Zoom® using an iPad®, and aim to get 120 minutes of aerobic activity and 30 minutes of strength exercises each week.
  In addition, they will attend in-person cooking classes-twice a month during the first 6 months and once a month for the next 12 months. In these 60-minute classes, instructors will teach cooking skills, and participants will practice on their own or with a partner, depending on their comfort level. They will learn how to safely use kitchen tools and appliances (like ovens, blenders, knives, and measuring cups) and prepare simple meals or snacks.
  Other Names: eSLD+Chef-ID
  Arms: Weight Loss Plus Cooking
Behavioral: Traditional Weight Loss — Participants in the eSLD group will follow a healthy eating plan using the enhanced stoplight diet, meet once a month with a health coach on Zoom® using an iPad®, and aim to get 120 minutes of aerobic activity and 30 minutes of strength exercises each week.
  They will also receive short (2-minute) video messages from their coach-twice a month during the first 6 months and once a month after that. These videos will include feedback on their progress, reminders about their goals, and tips to help them stay on track with healthy eating and exercise.
  Other Names: eSLD
  Arms: Traditional Weight Loss

SUMMARY:
The goal of this study is to see if adding hands-on cooking classes to a weight management program (called Chef-ID) helps young adults with intellectual disabilities lose more weight and keep it off compared to a standard weight loss program. The study will last 24 months and include three phases: 6 months of active support, 12 months of maintenance, and 6 months with no contact.

The investigators will look at how much weight participants lose over the first 18 months. Changes in cooking skills, body fat, health markers (like blood pressure and cholesterol), daily living skills, and caregiver stress will be tracked. Finally, factors that might help or prevent weight loss, and how changes in weight and body fat are linked to overall health will be explored.

This research will help inform on how to better support healthy lifestyles for people with intellectual disabilities.

DETAILED DESCRIPTION:
This study will compare two different approaches to long-term weight loss in young adults (ages 18-30) with mild-to-moderate intellectual disabilities. One group will follow a traditional weight loss program (called eSLD), while the other will follow the same program plus take part in in-person cooking classes (called eSLD+Chef-ID). A total of 114 participants will be randomly assigned by computer to one of the two groups for a 24-month study, which includes 6 months of active support, 12 months of follow-up, and 6 months with no contact.

All participants will follow a simple diet called the "enhanced stoplight diet" and try to get at least 120 minutes of aerobic exercise and 30 minutes of strength training each week. Participants be given an iPad® with pre-recorded exercise videos, a wearable fitness tracker, and will have monthly Zoom check-ins with a health coach for 18 months.

Those in the eSLD+Chef-ID group will also attend fun, hands-on cooking classes twice a month during the first 6 months and once a month from months 7-18. Participants in the traditional eSLD group will receive short motivational video messages from their coach instead of cooking classes.

Weight will be measured at the beginning, 6, 12, 18, and 24 months. Other health measures like cooking skills, body fat, blood pressure, and caregiver stress will also be collected during lab and home visits. The goal is to find out whether learning to cook helps improve long-term weight loss and overall health in this community.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of mild-to-moderate intellectual disability (ID).
2. 18-35 years of age.
3. BMI >24.9, Body weight <350lbs.
4. Sufficient functional ability to understand directions, communicate preferences, e.g., foods, wants, and can communicate through spoken language e.g., request more to eat/drink, asks for assistance with food preparation.
5. Living at home with a parent/guardian, or in a supported living environment with a caregiver who assists with food shopping, meal planning, and meal preparation and agrees to serve as a study partner.
6. Plan to attend all study required visits over the next 24 mos.

Exclusion Criteria:

1. Unable to participate in PA.
2. Insulin dependent diabetes as this condition requires medical monitoring beyond the scope of this study.
3. Participation in a weight management program involving diet, PA, or pharmacotherapy in the past 6 mos.
4. Diagnosis of Prader-Willi Syndrome.
5. Pregnancy during the previous 6 mos., currently lactating or planned pregnancy in the following 24 mos. Participants who become pregnant will be removed from the study and referred to appropriate agencies for consultation.
6. Serious medical risk, e.g., cancer, recent heart attack, stroke, angioplasty as determined by the PCP.
7. Unwilling to be randomized.
8. Unable to participate in small group, in-person instruction.
9. Use of wheelchair or power chair as primary locomotion.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Weight Loss Between Arms | Baseline to 18 months
  Weight will be measured in duplicate on a calibrated scale after an overnight fast during a laboratory visit at baseline, 6, 12, and 18 mos.

SECONDARY OUTCOMES:
Changes in Weight | Baseline to 24 months
  Weight will be measured in duplicate on a calibrated scale during a laboratory visit after an overnight fast at baseline, 6, 12, and 18 mos and during a home visit at 24 mos.
Activities of Daily Living | Baseline to 24 months
  Activities of Daily Living will be assessed using the 17-item Waisman Activities of Daily Living survey, which was specifically developed for and validated in adolescents and adults with intellectual disabilities. Scores range from 0 to 34, with a higher score indicating increased independence.
Caregiver Strain | Baseline to 24 months
  Caregiver strain will be assessed using the Modified Caregiver Strain Index which measures caregivers' levels of strain, a combination of stress and burden. The index assesses 13 aspects of physical health, family finances, social interactions, time demands, and employment. Scores range from 0 to 26, with a higher score indicating increased caregiver strain.
Fat Mass | Baseline to 18 months
  Body composition will be assessed using dual energy x-ray absorptiometry (DXA -Prodigy Advance Plus, GE, Madison WI). Pregnancy testing will be completed by all females prior to each DXA test. All participants will wear a hospital gown during DXA scans to standardize clothing.
Fat-free Mass | Baseline to 18 months
  Body composition will be assessed using dual energy x-ray absorptiometry (DXA -Prodigy Advance Plus, GE, Madison WI). Pregnancy testing will be completed by all females prior to each DXA test. All participants will wear a hospital gown during DXA scans to standardize clothing.
Percent Body Fat | Baseline to 18 months
  Body composition will be assessed using dual energy x-ray absorptiometry (DXA -Prodigy Advance Plus, GE, Madison WI). Pregnancy testing will be completed by all females prior to each DXA test. All participants will wear a hospital gown during DXA scans to standardize clothing.
High-density Lipoprotein (HDL) | Baseline to 18 months
  Whole blood will be drawn by a trained phlebotomist following a minimum 12-hr. fast and sent to The University of Kansas Health Systems for analysis.
Low-density Lipoprotein (LDL) | Baseline to 18 months
  Whole blood will be drawn by a trained phlebotomist following a minimum 12-hr. fast and sent to The University of Kansas Health Systems for analysis.
Fasting Glucose | Baseline to 18 months
  Whole blood will be drawn by a trained phlebotomist following a minimum 12-hr. fast and sent to The University of Kansas Health Systems for analysis.
Hemoglobin A1c (HbA1c) | Baseline to 18 months
  Whole blood will be drawn by a trained phlebotomist following a minimum 12-hr. fast and sent to The University of Kansas Health Systems for analysis.
Resting Blood Pressure | Baseline to 18 months
  Resting systolic and diastolic blood pressure will be measured on the non-dominant arm with participants seated in a chair and both feet flat on the ground.
Cooking Skills | Baseline to 18 months
  Cooking skills will be assessed using the Assessment of Functional Living Skills (AFLS): Independent Living Skills. Scores range from 48 to 336, with a lower score indicating increased independence.

OTHER OUTCOMES:
Skin Carotenoid Content | Baseline to 18 months
  We will assess skin carotenoid content with a finger scan using the Veggie Meter (Longevity Link Corporation), as biomarker of fruit and vegetables intake.
Dietary Intake | Baseline to 18 months
  Dietary intake will be assessed using the NHANES Dietary Screener Questionnaire which is a 26 item questionnaire that asks about the past months consumption of fruits, vegetables, dairy, added sugars, whole grains, red meat and processed meat. Based on the self-reported consumption, values for average daily intake are provided.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No